CLINICAL TRIAL: NCT06800079
Title: The Influence of Elastic Band Resistance Training on Knee Joint Muscle Strength and Performance-Related Parameters in Female Football Players: a Comparison of Three Development Phases
Brief Title: Elastic Band Training Effects on Knee Strength and Performance in Female Football Players
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Henrique Sousa (Other)
Collaborators: University Institute of Maia (Other); Portugal Football School, Federação Portuguesa de Futebol (Unknown)
Responsible Party: Sponsor-Investigator, Henrique Sousa, Henrique Sousa, MsC., University Institute of Maia
Organization: University Institute of Maia (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: EBT_HS_02
Record Dates: First submitted 2025-01-18; First posted 2025-01-29 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Physical Performance Parameters
Keywords: Elastic Bands; Resistance Training; Women; Football; Performance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental: Elastic Band Group (Experimental): Athletes that will participate in a bi-weekly elastic band resistance training program.
  Interventions: Other: EBT
- Control: Standard Group (No Intervention): Athletes that will continue doing their standard training regiment.

INTERVENTIONS:
Other: EBT — Elastic Band Resistance Training
  Arms: Experimental: Elastic Band Group

SUMMARY:
The goal of this clinical trial is to assess the effects of an 8-week strength training program with elastic bands on several physical components in female football players at the U15, U19, and Senior levels. The main question it aims to answer is:

Will a specific elastic band resistance training help improve some components of physical performance in female football players?

Participants will perform a bi-weekly elastic band resistance training program lasting 20 minutes per session over 8 weeks. This program will be incorporated into their in-season regimen, with assessments conducted in the week prior (week 0) and after the intervention (week 9).

DETAILED DESCRIPTION:
This study will involve U15´, U19´ and adult female football (soccer) players doing a specific elastic band training plan over a period of 8 weeks. This plan will be done twice a week and will consist of 6 exercises, divided into two training sessions, each lasting approximately 20 minutes.

The week before the study begins (week 0), a demonstration will be given of the assessments and training plan that will be carried out during the following weeks, so that the participants have a better idea of what will happen. In addition, their height and weight will also have to be measured, followed by the first assessments. They will also fill in a questionnaire about their training habits and injury history.

They will then be randomized into two possible groups: the experimental group (EG) and the control group (CG). If the participant stays in the EG, she will have to do the above protocol and if she stays in the CG, she will only have to do the assessments, which will be done in the familiarization week (week 0) and the ninth week (week 9).

ELIGIBILITY:
Inclusion Criteria:

* belong to the U-15, U-19 or Senior level of a women's football (soccer) club;
* be apart of a football championship (district or national)

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-01-29 (Estimated); Primary Completion 2025-04-11 (Estimated); Study Completion 2025-04-28 (Estimated)

PRIMARY OUTCOMES:
Knee extension and flexion isometric strength | The evaluations will be conducted in the week prior (week 0) and after the intervention (week 9).
  Maximal isometric knee extension and flexion force will be measured using a handheld dynamometer (DynaMo Plus, VALD Performance, Brisbane, Queensland, Australia). For the knee extension assessment, participants will be in a seated position, whereas during the knee flexion evaluation, the participants will be in a prone position. To generate their maximal torque, the dynamometer chain length will be adjusted so that their knee angle will be at ∼60° and ∼30°, for the knee extension and flexion, respectively. Participants will then apply a maximal isometric effort, maintaining it for 5s, without any subsidiary body movements.
Vertical jump | The evaluations will be conducted in the week prior (week 0) and after the intervention (week 9).
  Jump height will be evaluated using force plates (ForceDecks, Vald). The players will perform the countermovement jump, where they will begin from an upright position; a rapid downward movement to a knee angle of ∼90°, immediately transitioning to propel themselves upwards into the air.
Change of direction sprint | The evaluations will be conducted in the week prior (week 0) and after the intervention (week 9).
  The Modified T-Test will be implemented to assess change of direction sprint. This evaluation has within itself directional changes such as forward sprinting, left and right-side shuffling, and backpedaling. Photocells (WhittyGate, Microgate, Bolzano, Italy) will be used for a more precise time count.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Maia, Maia, Porto District, Portugal

IPD SHARING:
Plan to Share IPD: Undecided